CLINICAL TRIAL: NCT04913818
Title: The Effects of the Buddy-Up Dyadic Physical Activity (BUDPA) Program on the Health Outcomes of Care Dyads of Dementia: A Pilot Feasibility Study
Brief Title: Effects of the Buddy-Up Dyadic Physical Activity Program on Health Outcomes of Care Dyads of Dementia: A Pilot Study
Acronym: BUDPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BUDPA
Record Dates: First submitted 2021-04-16; First posted 2021-06-04 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Mild Dementia; Moderate Dementia
Keywords: mild to early moderate dementia

STUDY DESIGN:
Intervention Model Description: To examine the feasibility and preliminary effect of a partnering exercise program on the health outcomes of the PwD and their family caregivers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUDPA Program (Experimental): The overall program includes 12 weekly 1-hour training class. Each session starts with a 10-minute warm-up period using stretching exercise and stationary mobilizing exercise for trunk and limb joints at both upper and lower bodies and followed by a session of four to six selected partnering exercise, with duration increase gradually from 20 minutes to 40 minutes in four weeks' time. The Borg Rate of Perceived Exertion (Borg RPE) will be used to monitor the exercise intensity. The research assistant will explain the Borg RPE scale to the subjects and instruct them to speed up or slow down their movements in order to achieve a feeling of 'somewhat hard' at the Borg RPE rating of 12-14. The training session will end with a 10-minute cool down exercise session.
  Interventions: Behavioral: BUDPA Program
- Usual Care (Active Comparator): Activities will be provided by the elderly community center such as dementia or caregiver supporting service. They will be allowed to use the regular service provided such services are not related to physical activity or exercise training.
  Interventions: Other: Control arm (Usual care)

INTERVENTIONS:
Behavioral: BUDPA Program — The overall program includes 12 weekly 1-hour training class. Each session starts with a 10-minute warm-up period using stretching exercise and stationary mobilizing exercise for trunk and limb joints at both upper and lower bodies (e.g. shoulders, elbows, wrists, hips, knees and ankles), and followed by a session of four to six selected partnering exercise, with duration increase gradually from 20 minutes to 40minutes in four weeks' time. The Borg Rate of Perceived Exertion (Borg RPE) will be used to monitor the exercise intensity. The Research assistant will explain the Borg RPE scale to the subjects and instruct them to speed up or slow down their movements. The training session will end with a 10-minute cool down session with walking exercise and stationary trunk and limb mobilizing exercise involving joints of shoulders, elbows, wrists, hips, knees, and ankles.
  Arms: BUDPA Program
Other: Control arm (Usual care) — Active Comparator: Usual Care Activities will be provided by the elderly community center such as dementia or caregiver supporting service. They will be allowed to use the regular service provided such services are not related to physical activity or exercise training
  Arms: Usual Care

SUMMARY:
This project seeks to develop a novel dyadic intervention (titled as Buddy-Up Dyadic Physical Activity; BUDPA), using exercise as the common treatment component to improve the cognitive outcomes of persons with dementia and manage the stress-related symptoms of their family caregivers.

DETAILED DESCRIPTION:
This project is a pilot study that seeks to develop a novel dyadic BUDPA intervention, using exercise as the common treatment component to improve the cognitive outcomes of persons with dementia and manage the stress-related symptoms of their family caregivers. BUDPA has integrated the concept of developing social capital for dementia management. By applying partner exercise, the longer-term provider for this therapeutic care will be shifted from service providers to the family caregivers and the persons with dementia. Helping them to translate the practice to a home-care setting further strengthens the notions of family responsibility and ability in dementia management. BUDPA fully engages the care dyads in a mutual helping relationship during the exercise training. The partner exercise also creates a platform to enable more meaningful encounter within the care dyad. The family caregivers are facilitated to find meaning in the caregiving process, which eventually can benefit their role commitment and mental wellness. Also, the use of mixed-method study design can provide high quality findings to inform both the feasibility and preliminary effects of the BUDPA program.

ELIGIBILITY:
Inclusion Criteria:

For PwD,

* confirmed diagnosed of mild to moderate-intensity dementia
* cognitive impairment as indicated by a HK-Montreal Cognitive Assessment (Hong Kong version; HK-MoCA) score of 8-19 to indicate mild to early moderate dementia will be recruited

For family caregivers

* live together with the PwD
* identify as the primary family caregivers of the PwD

Exclusion Criteria:

* engaging in > 60 minutes per week of moderate or more vigorous exercise in the previous six months
* acute muscular-skeletal problem, stroke or cardio-respiratory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | Baseline
  evaluating various domains (i.e. attention and working memory, episodic memory, complex attention, executive function and task switching) of cognition of the PwD
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 6th week
  evaluating various domains (i.e. attention and working memory, episodic memory, complex attention, executive function and task switching) of cognition of the PwD
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 12th week
  evaluating various domains (i.e. attention and working memory, episodic memory, complex attention, executive function and task switching) of cognition of the PwD
Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-Cog) | 18th week
  evaluating various domains (i.e. attention and working memory, episodic memory, complex attention, executive function and task switching) of cognition of the PwD
Zarit Burden Interview (Chinese version; ZBI-C) | Baseline
  measuring the caregiving burden of the family caregivers
Zarit Burden Interview (Chinese version; ZBI-C) | 6th week
  measuring the caregiving burden of the family caregivers
Zarit Burden Interview (Chinese version; ZBI-C) | 12th week
  measuring the caregiving burden of the family caregivers
Zarit Burden Interview (Chinese version; ZBI-C) | 18th week
  measuring the caregiving burden of the family caregivers

SECONDARY OUTCOMES:
Neuro-psychiatric Inventory (CNPI; Chinese version) | Baseline
  Evaluating neuro-psychiatric symptoms of the PwD
Neuro-psychiatric Inventory (CNPI; Chinese version) | 6th week
  Evaluating neuro-psychiatric symptoms of the PwD
Neuro-psychiatric Inventory (CNPI; Chinese version) | 12th week
  Evaluating neuro-psychiatric symptoms of the PwD
Neuro-psychiatric Inventory (CNPI; Chinese version) | 18th week
  Evaluating neuro-psychiatric symptoms of the PwD
Lawton Instrumental activities of daily living IADL(IADL) Questionnaire | Baseline
  Measuring the ability of engaging in instrumental Activities of daily living(ADL) for the Pwd
Lawton Instrumental activities of daily living IADL(IADL) Questionnaire | 6th week
  Measuring the ability of engaging in instrumental Activities of daily living(ADL) for the Pwd
Lawton Instrumental activities of daily living IADL(IADL) Questionnaire | 12th week
  Measuring the ability of engaging in instrumental Activities of daily living(ADL) for the Pwd
Lawton Instrumental activities of daily living IADL(IADL) Questionnaire | 18th week
  Measuring the ability of engaging in instrumental Activities of daily living(ADL) for the Pwd
Profile of Mood State (Abbreviated) | Baseline
  Measuring the six identifiable mood status including tension anxiety, depression dejection, anger hostility, vigor activity, fatigue inertia and confusion bewilderment of family caregivers
Profile of Mood State (Abbreviated) | 6th week
  Measuring the six identifiable mood status including tension anxiety, depression dejection, anger hostility, vigor activity, fatigue inertia and confusion bewilderment of family caregivers
Profile of Mood State (Abbreviated) | 12th week
  Measuring the six identifiable mood status including tension anxiety, depression dejection, anger hostility, vigor activity, fatigue inertia and confusion bewilderment of family caregivers
Profile of Mood State (Abbreviated) | 18th week
  Measuring the six identifiable mood status including tension anxiety, depression dejection, anger hostility, vigor activity, fatigue inertia and confusion bewilderment of family caregivers
Positive Affect Index | Baseline
  Assessing the current relationship quality of family caregivers with PwD. It covers the feelings of understanding, trust, respect, fairness and affection.
Positive Affect Index | 6th week
  Assessing the current relationship quality of family caregivers with PwD. It covers the feelings of understanding, trust, respect, fairness and affection.
Positive Affect Index | 12th week
  Assessing the current relationship quality of family caregivers with PwD. It covers the feelings of understanding, trust, respect, fairness and affection.
Positive Affect Index | 18th week
  Assessing the current relationship quality of family caregivers with PwD. It covers the feelings of understanding, trust, respect, fairness and affection.
Positive Aspects of Caregiving Scale | Baseline
  To measure caregiver gain of the family caregivers. It measures two components, self-affirmation and outlook on life.
Positive Aspects of Caregiving Scale | 6th week
  To measure caregiver gain of the family caregivers. It measures two components, self-affirmation and outlook on life.
Positive Aspects of Caregiving Scale | 12th week
  To measure caregiver gain of the family caregivers. It measures two components, self-affirmation and outlook on life.
Positive Aspects of Caregiving Scale | 18th week
  To measure caregiver gain of the family caregivers. It measures two components, self-affirmation and outlook on life.

CONTACTS AND LOCATIONS:
Overall Officials: Doris, Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.

REFERENCES:
- [Background] Dassel KB, Carr DC. Does Dementia Caregiving Accelerate Frailty? Findings From the Health and Retirement Study. Gerontologist. 2016 Jun;56(3):444-50. doi: 10.1093/geront/gnu078. Epub 2014 Aug 26. PMID 25161263
- [Background] Van't Leven N, Prick AE, Groenewoud JG, Roelofs PD, de Lange J, Pot AM. Dyadic interventions for community-dwelling people with dementia and their family caregivers: a systematic review. Int Psychogeriatr. 2013 Oct;25(10):1581-603. doi: 10.1017/S1041610213000860. Epub 2013 Jul 24. PMID 23883489
- [Background] Yu DSF, Cheng ST, Wang J. Unravelling positive aspects of caregiving in dementia: An integrative review of research literature. Int J Nurs Stud. 2018 Mar;79:1-26. doi: 10.1016/j.ijnurstu.2017.10.008. Epub 2017 Oct 16. PMID 29128685
- [Background] Hernandez SS, Sandreschi PF, da Silva FC, Arancibia BA, da Silva R, Gutierres PJ, Andrade A. What are the Benefits of Exercise for Alzheimer's Disease? A Systematic Review of the Past 10 Years. J Aging Phys Act. 2015 Oct;23(4):659-68. doi: 10.1123/japa.2014-0180. Epub 2014 Nov 21. PMID 25414947
- [Background] Puterman E, Weiss J, Lin J, Schilf S, Slusher AL, Johansen KL, Epel ES. Aerobic exercise lengthens telomeres and reduces stress in family caregivers: A randomized controlled trial - Curt Richter Award Paper 2018. Psychoneuroendocrinology. 2018 Dec;98:245-252. doi: 10.1016/j.psyneuen.2018.08.002. Epub 2018 Aug 2. PMID 30266522
- [Background] Prick AE, de Lange J, Scherder E, Twisk J, Pot AM. The effects of a multicomponent dyadic intervention on the mood, behavior, and physical health of people with dementia: a randomized controlled trial. Clin Interv Aging. 2016 Mar 31;11:383-95. doi: 10.2147/CIA.S95789. eCollection 2016. PMID 27099480
- [Background] Gellert P, Ziegelmann JP, Warner LM, Schwarzer R. Physical activity intervention in older adults: does a participating partner make a difference? Eur J Ageing. 2011 Jul 7;8(3):211. doi: 10.1007/s10433-011-0193-5. eCollection 2011 Sep. PMID 28798651
- [Background] Yeung PY, Wong LL, Chan CC, Leung JL, Yung CY. A validation study of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) in Chinese older adults in Hong Kong. Hong Kong Med J. 2014 Dec;20(6):504-10. doi: 10.12809/hkmj144219. Epub 2014 Aug 15. PMID 25125421
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Chu LW, Chiu KC, Hui SL, Yu GK, Tsui WJ, Lee PW. The reliability and validity of the Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) among the elderly Chinese in Hong Kong. Ann Acad Med Singap. 2000 Jul;29(4):474-85. PMID 11056778
- [Background] Leung VP, Lam LC, Chiu HF, Cummings JL, Chen QL. Validation study of the Chinese version of the neuropsychiatric inventory (CNPI). Int J Geriatr Psychiatry. 2001 Aug;16(8):789-93. doi: 10.1002/gps.427. PMID 11536346
- [Background] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Background] Chen KM, Snyder M, Krichbaum K. Translation and equivalence: the Profile of Mood States Short Form in English and Chinese. Int J Nurs Stud. 2002 Aug;39(6):619-24. doi: 10.1016/s0020-7489(01)00068-2. PMID 12100873
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- See also: Alzheimer's Disease International. World Alzheimer Report-2015 — https://www.alz.co.uk/research/world-report-2015
- See also: Alzheimer's Disease International. World Alzheimer Report-2016 — https://www.alz.co.uk/research/world-report-2016
- See also: World Health Organization. Dementia: A public health priority — https://www.who.int/publications/i/item/dementia-a-public-health-priority

DOCUMENTS (1):
  • Informed Consent Form (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04913818/ICF_000.pdf